CLINICAL TRIAL: NCT04859504
Title: Dual-channel Transcranial Alternating Current Stimulations Targeting Negative Symptoms in Schizophrenia Patients: a Randomized Clinical Trial
Brief Title: Developing Dual-channel Transcranial Alternating Current Stimulations Targeting Negative Symptoms in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20191836
Record Dates: First submitted 2021-04-01; First posted 2021-04-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Transcranial Alternating Current Stimulations; Negative Symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tACS (Active Comparator): Active tACS will be applied twice daily for 5 days. In each session, dual-channel high-density theta(7Hz) tACS stimulations will be delivered over the right DLPFC (one anodal electrode at F4, between -1.2mA and 1.2 mA; two cathodal electrodes at AF4 and FC6, between -0.6mA and 0.6mA) and cerebellum (one anodal electrode at Oz, between -1 mA and 1mA; two cathodal electrodes at PO3 and PO4, between -0.5mA and 0.5mA) lasting 20 minutes.
  Interventions: Device: transcranial alternating current stimulation (NE Starstim)
- Sham tACS (Sham Comparator): Sham tACS will be also applied twice daily for 5 days.The parameters of tACS electrodes numbers, locations, and current duration are all the same with active tACS. But sham tACS begin with a fade in over 3s to the peak, followed immediately by no current stimulation for 20 minutes and a fade out of 3s.
  Interventions: Device: transcranial alternating current stimulation (NE Starstim)

INTERVENTIONS:
Device: transcranial alternating current stimulation (NE Starstim) — dual-channel theta-tACS over right DLPFC and cerebellum simultaneously

SUMMARY:
Negative symptoms are core symptoms in schizophrenia which play an important role in clinical outcomes and impede patients to return to society. Anti-psychotic medicines have shown limited effect in improving negative symptoms and cognitive functioning, whereas non-invasive neuromodulations, i.e. , transcranial alternating current stimulation (tACS), have shown promising potentials. Recently new evidence of brain structural and functional alterations has been provided by neuroimaging studies. Brady RO et al. found cerebellar-prefrontal network connectivity was related to negative symptoms in schizophrenia. It provides clues for developing a new tACS protocol targeting improving negative symptoms, in which dual-channel high-density alternating current stimulations were delivered over both the right dorsolateral prefrontal cortex and cerebellum simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* meet the DSM-V diagnostic criteria for schizophrenia;
* present with prominent negative symptoms with PANSS-negative scores >20, at least one score of PANSS N1-N7 >3, and reductive ratio of PANSS-negative in the past two weeks before recruitment <10%;
* stable usage and dosage of anti-psychotic medicines in the past two weeks and during the tACS intervention.
* age within 18-60;
* illness duration >1year;
* education at least 6 years;
* written consent of receiving tACS intervention.

Exclusion Criteria:

* Meet any DSM-V diagnostic criteria of any other psychiatric disorders besides schizophrenia ;
* any history of alcohol or substance dependence in the past 3 months;
* any other major physical disease (i.e., Sensorimotor disorder, neurological disease);
* any metal implants or any other tACS contraindication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
reductive ratio of PANSS-negative symptoms scores | At 1 week and 3 weeks
  differences of reductive ratio of PANSS-negative symptoms scores after between active and sham tACS

SECONDARY OUTCOMES:
changes of PANSS total scores | At 1 week and 3 weeks
  changes of PANSS total scores before and after active or sham tACS
cognitive functioning changes using MCCB | At 1 week and 3 weeks
  changes of MCCB scores before and after active or sham tACS
changes of P300 activity | At 1 week
  changes of P300 activity at baseline and after 10-session tACS
changes of MMN activity | At 1 week
  changes of MMN activity at baseline and after 10-session tACS
changes of power of resting-state EEG activity | At 1 day and 1 week
  changes of power of resting-state EEG activity at baseline, after 1-session tACS and after 10-session tACS
centroid value from fNIRS recording before and after active or sham tACS | At 1 week
  centroid value from fNIRS recording before and after active or sham tACS
Integral value from fNIRS recording before and after active or sham tACS | At 1 week
  Intergral value from fNIRS recording before and after active or sham tACS

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Tang, PhD, Principal Investigator — Shanghai Mental Health Center; Jianhua Sheng, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (2):
- China (2):
  - Zhengjiang Mental Health Center, Zhenjiang, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
We will decide IPD or not when the clinical trial is completed.

REFERENCES:
- [Background] Brady RO Jr, Gonsalvez I, Lee I, Ongur D, Seidman LJ, Schmahmann JD, Eack SM, Keshavan MS, Pascual-Leone A, Halko MA. Cerebellar-Prefrontal Network Connectivity and Negative Symptoms in Schizophrenia. Am J Psychiatry. 2019 Jul 1;176(7):512-520. doi: 10.1176/appi.ajp.2018.18040429. Epub 2019 Jan 30. PMID 30696271
- [Background] Reinhart RMG, Nguyen JA. Working memory revived in older adults by synchronizing rhythmic brain circuits. Nat Neurosci. 2019 May;22(5):820-827. doi: 10.1038/s41593-019-0371-x. Epub 2019 Apr 8. PMID 30962628
- [Background] Smith RC, Md WL, Wang Y, Jiang J, Wang J, Szabo V, Faull R, Jin H, Davis JM, Li C. Effects of transcranial direct current stimulation on cognition and symptoms in Chinese patients with schizophrenia✰. Psychiatry Res. 2020 Feb;284:112617. doi: 10.1016/j.psychres.2019.112617. Epub 2019 Nov 2. PMID 31806403